CLINICAL TRIAL: NCT02124772
Title: An Open-Label, Dose-Escalation, Phase I/II Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of the MEK Inhibitor Trametinib in Children and Adolescents Subjects With Cancer or Plexiform Neurofibromas and Trametinib in Combination With Dabrafenib in Children and Adolescents With Cancers Harboring V600 Mutations
Brief Title: Study to Investigate Safety, Pharmacokinetic (PK), Pharmacodynamic (PD) and Clinical Activity of Trametinib in Subjects With Cancer or Plexiform Neurofibromas and Trametinib in Combination With Dabrafenib in Subjects With Cancers Harboring V600 Mutations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116540; 2013-003596-35 (EudraCT Number); CTMT212X2101 (Other: Novartis)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Cancer
Keywords: v600-mutation; neuroblastoma; Trametinib; pediatrics; Langerhans Cell Histiocytosis; low grade glioma; plexiform neurofibromas
MeSH Terms: conditions — Neoplasms; Neuroblastoma; Histiocytosis, Langerhans-Cell; Neurofibroma, Plexiform | interventions — trametinib; dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part A - TMT 0.0125 mg/kg/day (Experimental): Participants treated with trametinib 0.0125 mg/kg/day
  Interventions: Drug: Trametinib
- Part A - TMT 0.025 mg/kg/day (Experimental): Participants treated with trametinib 0.025 mg/kg/day
  Interventions: Drug: Trametinib
- Part A - TMT 0.032 mg/kg/day (Experimental): Participants under 6 years of age treated with trametinib 0.032 mg/kg/day
  Interventions: Drug: Trametinib
- Part A - TMT 0.04 mg/kg/day (Experimental): Participants treated with trametinib 0.04 mg/kg/day
  Interventions: Drug: Trametinib
- Part B - Neuroblastoma (Experimental): Participants with refractory or relapsed neuroblastoma treated with trametinib 0.025 mg/kg/day
  Interventions: Drug: Trametinib
- Part B - LGG fusion (Experimental): Participants with refractory or relapsed neuroblastoma treated with trametinib 0.025 mg/kg/day
  Interventions: Drug: Trametinib
- Part B - NF-1 with PN (Experimental): Participants with neurofibromatosis Type -1 associated plexiform neurofibromas (NF-1 with PN) treated with trametinib 0.025 mg/kg/day
  Interventions: Drug: Trametinib
- Part B - BRAF V600 mutant solid tumor (Experimental): Participants with BRAF V600 mutant solid tumors treated with trametinib 0.025 mg/kg/day
  Interventions: Drug: Trametinib
- Part C - TMT 0.025 mg/kg/day + 50% DRB RP2D (Experimental): Participants treated with a combination therapy of trametinib (0.025 mg/kg/day) plus 50% of the recommended phase II dose (RP2D) of dabrafenib monotherapy (2.63 mg/kg/day for <12 years old subjects and 2.25 mg/kg/day for ≥12 years old subjects)
  Interventions: Drug: Trametinib; Drug: Dabrafenib
- Part C - TMT 0.025 mg/kg/day + 100% DRB RP2D (Experimental): Participants treated with a combination therapy of trametinib (0.025 mg/kg/day) plus 100% of the recommended phase II dose (RP2D) of dabrafenib monotherapy (5.25 mg/kg/day for <12 years old subjects and 4.5 mg/kg/day for ≥12 years old subjects)
  Interventions: Drug: Trametinib; Drug: Dabrafenib
- Part C - TMT 0.032 mg/kg/day + 100% DRB RP2D (Experimental): Participants under 6 years of age treated with a combination therapy of trametinib (0.032 mg/kg/day) with 100% of the recommended phase II dose (RP2D) of dabrafenib monotherapy (5.25 mg/kg/day)
  Interventions: Drug: Trametinib; Drug: Dabrafenib
- Part D - LGG (Experimental): Participants with low grade glioma (LGG) treated with a combination therapy of trametinib (0.032 mg/kg/day for < 6 years old subjects and 0.025 mg/kg/day for ≥ 6 years old subjects) plus 100% of the recommended phase II dose (RP2D) of dabrafenib monotherapy (5.25 mg/kg/day for <12 years old subjects and 4.5 mg/kg/day for ≥12 years old subjects)
  Interventions: Drug: Trametinib; Drug: Dabrafenib
- Part D - LCH (Experimental): Participants with Langerhans cell histiocytosis (LCH) treated with a combination therapy of trametinib (0.032 mg/kg/day for < 6 years old subjects and 0.025 mg/kg/day for ≥ 6 years old subjects) plus 100% of the recommended phase II dose (RP2D) of dabrafenib monotherapy (5.25 mg/kg/day for <12 years old subjects and 4.5 mg/kg/day for ≥12 years old subjects)
  Interventions: Drug: Trametinib; Drug: Dabrafenib

INTERVENTIONS:
Drug: Trametinib — Trametinib was administered orally, once daily. It was available in tablets (0.125 mg, 0.5 mg, 2 mg dose) as well as in powder form for oral solution (0.05 mg/mL dose).
Drug: Dabrafenib — Dabrafenib was administered orally, twice daily. The daily dose was divided into two equal doses. It was available in capsules (50 mg and 75 mg), dispersible tablets (10 mg) and powder for oral suspension (10 mg/mL dose).
  Arms: Part C - TMT 0.025 mg/kg/day + 100% DRB RP2D; Part C - TMT 0.025 mg/kg/day + 50% DRB RP2D; Part C - TMT 0.032 mg/kg/day + 100% DRB RP2D; Part D - LCH; Part D - LGG

SUMMARY:
This was a 4-part (Part A, Part B, Part C and Part D), Phase I/IIa, multi-center, open label, study in pediatric subjects with refractory or recurrent tumors.

Part A was a repeat dose, dose escalation and expansion phase that identified the recommended phase II dose (RP2D) of trametinib monotherapy. Part B evaluated the preliminary activity of trametinib monotherapy in 4 disease-specific cohorts of subjects. Part C was aimed to determine the safety, tolerability and preliminary activity of the RP2D of trametinib in combination with a limited dose escalation of dabrafenib. Part D evaluated the preliminary activity of trametinib in combination with dabrafenib in 2 disease-specific cohorts of subjects.

The overall goal of this trial was to efficiently establish safe, pharmacologically relevant dose of trametinib monotherapy and trametinib in combination with dabrafenib in infants, children and adolescents and determine preliminary activity of trametinib monotherapy and trametinib in combination with dabrafenib in selected recurrent, refractory or unresectable childhood tumors.

DETAILED DESCRIPTION:
This was a 4-part (Part A, Part B, Part C and Part D), Phase I/IIa, multi-center, open label, study in pediatric subjects with refractory or recurrent tumors.

Part A was a repeat dose, dose escalation and expansion phase that identified the recommended phase II dose (RP2D) of trametinib monotherapy using a 3 + 3 dose- escalation procedure. The starting dose level of trametinib was 0.0125 mg/kg/day, the second dose level was 0.025 mg/kg/day and the third dose level was 0.040 mg/kg/day. Additionally, in Part A extension an intermediate trametinib dose level of 0.032 mg/kg/day was assessed in subjects under 6 years of age. In all cohorts, the total daily trametinib dose was not to exceed the adult dose (2 mg) in any subject.

Part B evaluated the preliminary activity of trametinib monotherapy in 4 disease-specific cohorts of subjects:

B1: Refractory or relapsed neuroblastoma B2: Recurrent or unresectable low grade glioma (LGG) with BRAF tandem duplication with fusion (glioma fusion) B3: Neurofibromatosis Type -1 associated plexiform neurofibromas (NF-1 with PN) that are unresectable and medically significant B4: BRAF V600 mutant tumors In Part B it was used the RP2D of trametinib (0.025 mg/kg/day) determined in Part A.

Part C was a 3+3 study design to determine the safety, tolerability and preliminary activity of the RP2D of trametinib in combination with a limited dose escalation of dabrafenib. The trametinib dose administered in Part C was based on the trametinib monotherapy RP2D from Part A (0.025 mg/kg/day). For the evaluation of combination therapy in this study, the starting dose of dabrafenib was 50% of the monotherapy RP2D established in a separate study: 2.63 mg/kg/day (<12 years old subjects) and 2.25 mg/kg/day (≥12 years old subjects). The second dose level of dabrafenib was 100% of the monotherapy RP2D: 5.25 mg/kg/day (<12 years old subjects) and 4.5 mg/kg/day (≥12 years old subjects).

Additionally, in Part C extension, the trametinib dose determined from Part A extension (0.032 mg/kg/day) with 100% pediatric RP2D of dabrafenib (5.25 mg/kg/day) was assessed in subjects under 6 years of age.

In all cohorts, the total daily trametinib dose was not to exceed the adult dose (2 mg) in any subject and the total daily dabrafenib dose was not to exceed the adult dose (300 mg) in any subject.

Part D evaluated the preliminary activity of trametinib in combination with dabrafenib in two disease-specific cohorts of subjects diagnosed with low grade glioma (LGG) and Langerhans cell histiocytosis (LCH).

In Part D it was used the RP2D of the combination treatment determined in Part C (0.025 mg/kg/day trametinib and the 100% RP2D of dabrafenib) in subjects 6 years to < 18 years of age. Additionally, once Part C extension had defined the trametinib RP2D for subjects under 6 years of age, this dose was used for the remaining subjects enrolled in Part D (0.032 mg/kg/day trametinib and the 100% RP2D of dabrafenib).

The overall goal of this trial was to efficiently establish safe, pharmacologically relevant dose of trametinib monotherapy and trametinib in combination with dabrafenib in infants, children and adolescents and determine preliminary activity of trametinib monotherapy and trametinib in combination with dabrafenib in selected recurrent, refractory or unresectable childhood tumors.

ELIGIBILITY:
Inclusion Criteria:

* General Eligibility Criteria (All Parts)
* Written informed consent - a signed informed consent and/or assent (as age appropriate) for study participation including PK sampling will be obtained according to institutional guidelines.
* Male or female between one month and <18 years of age (inclusive) at the time of signing the informed consent form (Part C and Part D between 12 months and <18 years of age, inclusive).
* Must have a disease that is relapsed/refractory to all potentially curative standard treatment regimens or must have a current disease for which there is no known curative therapy, or therapy proven to prolong survival with an acceptable quality of life.
* Prior therapy: The subject's disease (i.e. cancer, neurofibromatosis type 1 [NF-1] with plexiform neurofibroma [PN], or Langerhans cell histocytosis [LCH]) must have relapsed after or failed to respond to frontline curative therapy or there must not be other potentially curative treatment options available. Curative therapy may include surgery, radiation therapy, chemotherapy, or any combination of these modalities. All subjects must have recovered to grade <=1 from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to enrollment. Prior therapy includes; myelosuppressive chemotherapy, differentiating agents/ biologic response modifiers (small molecules, antibodies, viral therapies) (anti-cancer agent), non-myelosuppressive anticancer agents, investigational agent, radiation therapy, stem cell transplantation or infusion, number of prior treatment regimens, colony stimulating factors, corticosteroids.
* Performance score of >=50% according to the Karnofsky/Lansky performance status scale.
* Females of child-bearing potential must be willing to practice acceptable methods of birth control. Additionally, females of childbearing potential must have a negative serum pregnancy test within 7 days prior to start of study drugs, throughout treatment period and for 4 months after last dose of study drugs.
* Must have adequate organ function as defined by the following values: renal function - 24 hr creatinine clearance (revised Schwartz formula), or radioisotope glomerular filtration rate (GFR) >=60 milliliter (mL) per minute per 1.73 meter square (mL/min/1.73m^2); or a serum creatinine <=upper limit of normal (ULN) for age and gender; liver functions as bilirubin (sum of conjugated + unconjugated) <=1.5 x ULN for age, alanine aminotransferase (ALT) <=2.5 x ULN; for the purposes of enrollment and toxicity monitoring the ULN for ALT will be 45 unit per liter (U/L); cardiac function - corrected QT (QTcB) interval <480 milliseconds (msec), left ventricular ejection fraction (LVEF) >=lower limit of normal (LLN) by ECHO.
* Able to swallow and retain enterally (per oral [PO] or nasogastric or gastric tube) administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Adequate Blood Pressure Control defined as: Blood pressure <= the 95th percentile for age, height, and gender.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.
* Specific Eligibility Criteria, Part A
* Subjects must meet general eligibility criteria.
* For the initial dose escalation to identify the maximum tolerable or PK target dose, age between 2 years and <18 years (inclusive) at the time of signing the informed consent form. Children < 2 years of age will be enrolled once the age specific expansion cohorts are open.
* Histologically confirmed solid tumors, which may include but are not limited to rhabdomyosarcoma and other soft tissue sarcomas, Ewing sarcoma family of tumors, osteosarcoma, neuroblastoma, Wilms' tumor, hepatic tumors, germ cell tumors, primary brain tumors, NF-1 associated PF and LCH. In subjects with brain stem gliomas the requirement for histological confirmation can be waived if a biopsy was not performed. For plexiform neurofibromas, histologic confirmation of tumor is not necessary in the presence of consistent clinical and radiological findings, but should be considered if malignant degeneration of a PN is clinically suspected.
* Measurable or evaluable tumors. Subjects with neuroblastoma that is only detectable by Meta-iodobenzylguanidine (MIBG) scan are eligible. Subjects with neuroblastoma that is only detected by bone marrow aspirate/biopsy or elevated homovanillic acid / vanillylmandelic acid (HVA/VMA) are not eligible.
* Adequate bone marrow function defined as absolute neutrophil count (ANC) >=1000/microliter, hemoglobin >=8.0 gram per deciliter (g/dL) (may receive red blood cell transfusions), platelets >=75,000/ microliter (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment).
* Specific Eligibility Criteria, Part B
* Subjects must meet general eligibility criteria. The specific eligibility criteria listed here will apply to subjects enrolling to different cohorts of Part B.
* Tumor tissue (archived or fresh) is required and must be available to be shipped to GSK or site specific laboratory.
* Solid tumor cohort (B1) specific criteria
* B1: Refractory or relapsed neuroblastoma
* B2: Recurrent or unresectable low grade gliomas with BRAF tandem duplication with fusion
* B3: Neurofibromatosis Type -1 associated plexiform neurofibromas (NF-1 with PN) that are unresectable and medically significant.
* B4: BRAF V600 mutant tumors.
* Specific Eligibility Criteria, Part C - Subjects must meet general eligibility criteria.
* Tumors that have been documented by CLIA or equivalent certified laboratory test to harbor BRAF V600 mutation at diagnosis or relapse
* Measurable or evaluable disease
* Adequate bone marrow function
* Specific Eligibility Criteria, Part D - Subjects must meet general eligibility criteria
* Measurable or evaluable disease
* Recurrent or refractory BRAFV600 mutant LGG or LCH tumors
* Adequate bone marrow function

Exclusion Criteria:

* Lactating or pregnant female.
* History of another malignancy including resected non-melanomatous skin cancer.
* Subjects with NF-1 associated optic pathway tumors are excluded if they are actively receiving therapy for the optic pathway tumor or do not meet criteria for PN or malignant solid tumor.
* Subjects with a history of NF-1 related cerebral vascular anomaly (such as Moyamoya).
* Subjects with NF-1 actively receiving therapy for the optic pathway tumor.
* Subjects with NF-1 and only PN lesions that cannot be evaluated by volumetric analysis (only applicable to Part B).
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Any prohibited medication(s), currently used or expected to be required.
* Any medications for treatment of left ventricular systolic dysfunction.
* Part B, Part C and Part D only: Previous treatment with dabrafenib or any BRAF inhibitor, trametinib or another MEK inhibitor, or and Extracellular signal-regulated kinase inhibitor (exception: prior treatment with sorafenib is permitted). Patients who have received prior dabrafenib or another BRAF inhibitor may enrol into Part B4. Patients who have had prior dabrafenib or BRAF inhibitor therapy may enroll in Part C or Part D if they have had prior benefit to dabrafenib or BRAF inhibitor monotherapy, as determined by the investigator.
* Administration of an investigational study treatment within 30 days preceding the first dose of study treatment(s) in this study.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study treatment or excipients that contraindicate their participation.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, or liver metastases).
* History of hepatic sinusoid obstructive syndrome (venoocculsive disease) within the prior 3 months.
* History of heparin-induced thrombocytopenia.
* History of interstitial lung disease or pneumonitis.
* History of or current evidence of retinal vein occlusion (RVO).
* For subjects with solid tumors that are not primary central nervous system (CNS) tumors or NF-1 associated plexiform neurofibromas subjects with symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression are excluded. NOTE: Subjects previously treated for these conditions that have had stable CNS disease (verified with consecutive imaging studies) for >3 months, are asymptomatic and are not currently taking corticosteroids, or are on stable dose or decreasing of corticosteroids for at least 7 days prior to enrolment are permitted.
* A history of known Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection. Subjects with laboratory evidence of cleared HBV and HCV infection may be enrolled.
* Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI CTCAE v4.0) Grade 2 or higher from previous anti-cancer therapy, except alopecia.
* Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption of drugs.
* A history or evidence of cardiovascular risk including: a QT interval corrected for heart rate using the Bazett's formula (QTcB) >=480 msec; a history or evidence of current clinically significant uncontrolled arrhythmias (clarification: Subjects with atrial fibrillation controlled for >30 days prior to dosing are eligible); a history of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization; a history or evidence of current >=Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines; subjects with intra-cardiac defibrillators; abnormal cardiac valve morphology (>=grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study. Subjects with prosthetic valves can be considered eligible provided they meet the criteria as stated above; Treatment refractory hypertension defined as a blood pressure of systolic >140 millimeter of mercury (mmHg) and/or diastolic >90 mmHg (or above 95th age-specific percentile listed in protocol), which cannot be controlled by anti-hypertensive therapy.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (10):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Memphis, Tennessee
- Novartis Investigative Site, Westmead, New South Wales, Australia
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- United Kingdom (2):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Whitlock JA, Geoerger B, Dunkel IJ, Roughton M, Choi J, Osterloh L, Russo M, Hargrave D. Dabrafenib, alone or in combination with trametinib, in BRAF V600-mutated pediatric Langerhans cell histiocytosis. Blood Adv. 2023 Aug 8;7(15):3806-3815. doi: 10.1182/bloodadvances.2022008414. PMID 36884302
- [Derived] Bouffet E, Geoerger B, Moertel C, Whitlock JA, Aerts I, Hargrave D, Osterloh L, Tan E, Choi J, Russo M, Fox E. Efficacy and Safety of Trametinib Monotherapy or in Combination With Dabrafenib in Pediatric BRAF V600-Mutant Low-Grade Glioma. J Clin Oncol. 2023 Jan 20;41(3):664-674. doi: 10.1200/JCO.22.01000. Epub 2022 Nov 14. PMID 36375115
- [Derived] Shahid S, Kushner BH, Modak S, Basu EM, Rubin EM, Gundem G, Papaemmanuil E, Roberts SS. Association of BRAF V600E mutations with vasoactive intestinal peptide syndrome in MYCN-amplified neuroblastoma. Pediatr Blood Cancer. 2021 Oct;68(10):e29265. doi: 10.1002/pbc.29265. Epub 2021 Jul 31. PMID 34331515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 16 investigative sites in 5 countries.
Pre-assignment Details: The participants were screened within 14 days prior to enrollment. After screening, the treatment period started on Cycle 1 Day 1.
Period: Overall Study
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH
Started | 3 | 19 | 12 | 16 | 11 | 10 | 10 | 10 | 3 | 9 | 6 | 20 | 10
Completed | 0 | 5 | 6 | 3 | 2 | 2 | 2 | 1 | 2 | 2 | 4 | 14 | 8
Not Completed | 3 | 14 | 6 | 13 | 9 | 8 | 8 | 9 | 1 | 7 | 2 | 6 | 2
Not completed — Lack of Efficacy | 2 | 0 | 0 | 1 | 2 | 3 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 4 | 1 | 5 | 2 | 1 | 1 | 5 | 0 | 3 | 1 | 3 | 1
Not completed — Withdrawal consent | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Investigator discretion | 0 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 7 | 2 | 5 | 4 | 3 | 4 | 1 | 1 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Total
Number analyzed (Participants) | 3 | 19 | 12 | 16 | 11 | 10 | 10 | 10 | 3 | 9 | 6 | 20 | 10 | 139
Age, Customized [Count of Participants; unit: Participants]
  < 2 years | 0 | 4 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 10
  2 - <6 years | 1 | 5 | 11 | 0 | 3 | 4 | 4 | 5 | 0 | 2 | 5 | 2 | 6 | 48
  6 - <12 years | 1 | 4 | 0 | 9 | 5 | 5 | 3 | 1 | 1 | 2 | 0 | 9 | 3 | 43
  ≥ 12 years | 1 | 6 | 0 | 5 | 2 | 1 | 2 | 4 | 2 | 5 | 0 | 9 | 1 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 6 | 7 | 6 | 5 | 5 | 5 | 0 | 6 | 4 | 10 | 2 | 64
  Male | 2 | 12 | 6 | 9 | 5 | 5 | 5 | 5 | 3 | 3 | 2 | 10 | 8 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 9
  White | 3 | 16 | 7 | 14 | 9 | 6 | 7 | 5 | 2 | 6 | 4 | 16 | 3 | 98
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 5 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 2 | 4 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events in Subjects Treated With Trametinib Monotherapy
Description: Incidence of treatment emergent adverse events is defined as number of participants with adverse events (AEs) and serious adverse events (SAEs), including changes from baseline in vital signs and laboratory results qualifying and reported as AEs. The number of participants in each category is reported in the table.
Time Frame: From the day of the first dose of trametinib up to 30 days after the last dose, up to maximum duration of 64 months
Population: All subjects who received at least one dose of trametinib in Part A and B
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor
Number analyzed (Participants) | 3 | 19 | 12 | 16 | 11 | 10 | 10 | 10
Participants
  AEs | 3 | 19 | 12 | 16 | 11 | 10 | 10 | 10
  Treatment-related AEs | 3 | 19 | 12 | 16 | 10 | 10 | 10 | 10
  SAEs | 1 | 8 | 3 | 11 | 6 | 6 | 6 | 5
  Treatment-related SAEs | 0 | 5 | 1 | 6 | 1 | 2 | 2 | 3
  Fatal SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs leading to discontinuation | 1 | 4 | 1 | 6 | 4 | 1 | 1 | 5
  AEs requiring dose interruptions | 0 | 12 | 6 | 14 | 3 | 8 | 5 | 8
  AEs requiring dose reductions | 0 | 9 | 5 | 9 | 2 | 4 | 3 | 7
  AEs requiring dose reductions or interruptions | 0 | 13 | 7 | 14 | 3 | 8 | 6 | 9

2. Primary Outcome: Average Steady State Plasma Concentration (Cavg) of Trametinib When Administered Alone (Monotherapy)
Description: Pharmacokinetic (PK) parameters were calculated based on trametinib plasma concentrations by using non-compartmental methods. The average steady state plasma concentration (Cavg) of trametinib was calculated as the ratio of area under the curve (AUC)/tau, where tau = 24 h for trametinib.
Time Frame: pre dose, 1, 2, 4, 7, 10 and 24 hours post trametinib dose on Cycle 1 Day 15. The duration of 1 cycle was 28 days.
Population: All subjects who received at least one dose of trametinib in Part A and B and provided an evaluable PK profile with a value for the outcome measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part B - All Tumor Types TMT 0.025 mg/kg/Day: Participants (all tumor types in Part B) treated with trametinib 0.025 mg/kg/day
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor | Part B - All Tumor Types TMT 0.025 mg/kg/Day
Number analyzed (Participants) | 3 | 18 | 9 | 15 | 9 | 10 | 10 | 9 | 38
ng/mL | 5.76 (24.8) | 13.9 (27.1) | 15.2 (16.9) | 21.3 (20.7) | 15.1 (36.0) | 13.2 (40.4) | 13.5 (25.1) | 15.8 (42.8) | 14.3 (35.8)

3. Secondary Outcome: Trough Concentration (Ctrough) of Trametinib When Administered Alone and in Combination With Dabrafenib
Description: Pharmacokinetic (PK) parameters were calculated based on trametinib plasma concentrations by using non-compartmental methods. Ctrough is defined as the observed plasma concentration just prior to the beginning of, or at the end, of a dosing interval.
Time Frame: pre dose on Cycle 1 Day 15. The duration of 1 cycle was 28 days.
Population: All subjects who received at least one dose of trametinib in Part A, B, C and D and provided an evaluable PK profile with a value for the outcome measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part B - LGG Fusion: Participants with recurrent or unresectable low grade glioma (LGG) with BRAF tandem duplication with fusion treated with trametinib 0.025 mg/kg/day
- Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D: Participants under 6 years of age (all tumor types in Part D) treated with a combination therapy of trametinib (0.032 mg/kg/day) with 100% of the recommended phase II dose (RP2D) of dabrafenib monotherapy (5.25 mg/kg/day)
- Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D: Participants (all tumor types in Part D) treated with a combination therapy of trametinib (0.025 mg/kg/day) plus 100% of the recommended phase II dose (RP2D) of dabrafenib monotherapy (5.25 mg/kg/day for <12 years old subjects and 4.5 mg/kg/day for ≥12 years old subjects)
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor | Part B - All Tumor Types TMT 0.025 mg/kg/Day | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 3 | 19 | 9 | 15 | 9 | 10 | 10 | 9 | 38 | 1 | 1 | 6 | 20 | 6 | 5 | 21
ng/mL | 4.37 (30.6) | 11.1 (44.0) | 10.2 (19.4) | 15.6 (30.1) | 10.7 (43.3) | 9.45 (53.6) | 9.25 (29.0) | 11.3 (50.3) | 10.1 (43.6) | 8.31 | 10.2 | 3.86 (34.9) | 8.60 (42.2) | 3.74 (66.3) | 3.05 (50.7) | 8.68 (38.6)

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Trametinib When Administered Alone and in Combination With Dabrafenib
Description: Pharmacokinetic (PK) parameters were calculated based on trametinib plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed plasma concentration following a dose.
Time Frame: pre dose, 1, 2, 4, 7, 10 and 24 hours post trametinib dose on Cycle 1 Day 15 (part A and B) and pre dose, 0.5, 1, 2, 3, 4, 6 and 8 hours post trametinib dose on Cycle 1 Day 15 (part C and D). The duration of 1 cycle was 28 days.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor | Part B - All Tumor Types TMT 0.025 mg/kg/Day | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 3 | 18 | 9 | 16 | 9 | 10 | 10 | 9 | 38 | 1 | 1 | 6 | 20 | 6 | 5 | 21
ng/mL | 9.61 (32.9) | 21.1 (33.3) | 26.1 (16.8) | 32.6 (28.9) | 26.6 (39.6) | 22.1 (41.9) | 21.6 (26.1) | 27.5 (31.6) | 24.2 (35.6) | 26.0 | 24.5 | 23.7 (36.3) | 22.9 (29.2) | 15.6 (52.5) | 25.9 (35.8) | 20.0 (38.1)

5. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Trametinib When Administered Alone and in Combination With Dabrafenib
Description: Pharmacokinetic (PK) parameters were calculated based on trametinib plasma concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) plasma concentration following a dose.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor | Part B - All Tumor Types TMT 0.025 mg/kg/Day | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 3 | 19 | 9 | 16 | 9 | 10 | 10 | 9 | 38 | 1 | 1 | 6 | 20 | 6 | 5 | 21
hours | 1.00 [1.00 to 2.00] | 2.00 [1.00 to 4.00] | 1.00 [1.00 to 2.00] | 2.00 [1.00 to 24.0] | 1.00 [1.00 to 4.00] | 1.50 [1.00 to 2.00] | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 1.50 [1.00 to 2.00] | 2.00 [1.00 to 3.00] | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 1.00] | 2.00 [1.00 to 4.00]

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast) of Trametinib When Administered Alone and in Combination With Dabrafenib
Description: Pharmacokinetic (PK) parameters were calculated based on trametinib plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for area under the curve calculation.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor | Part B - All Tumor Types TMT 0.025 mg/kg/Day | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 3 | 19 | 9 | 16 | 9 | 10 | 10 | 9 | 38 | 1 | 1 | 6 | 20 | 6 | 5 | 21
hours*ng/mL | 138 (24.8) | 341 (28.3) | 364 (16.9) | 413 (76.2) | 362 (36.0) | 316 (40.4) | 304 (36.9) | 379 (42.8) | 337 (38.6) | 290 | 331 | 122 (29.0) | 270 (35.8) | 118 (53.4) | 126 (30.7) | 255 (49.2)

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau at Steady-state (AUCtau) of Trametinib When Administered Alone and in Combination With Dabrafenib
Description: Pharmacokinetic (PK) parameters were calculated based on trametinib plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for area under the curve calculation. The duration of the dosing interval (tau) was 24 hours for trametinib.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor | Part B - All Tumor Types TMT 0.025 mg/kg/Day | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 3 | 18 | 9 | 15 | 9 | 10 | 10 | 9 | 38 | 1 | 1 | 6 | 20 | 6 | 5 | 21
hours*ng/mL | 138 (24.8) | 334 (27.1) | 364 (16.9) | 511 (20.7) | 362 (36.0) | 316 (40.4) | 323 (25.1) | 379 (42.8) | 343 (35.8) | 290 | 331 | 236 (28.4) | 308 (20.0) | 186 (23.7) | 228 (33.1) | 286 (28.4)

8. Secondary Outcome: Apparent Plasma Clearance (CL/F) of Trametinib When Administered Alone and in Combination With Dabrafenib
Description: Pharmacokinetic (PK) parameters were calculated based on trametinib plasma concentrations by using non-compartmental methods. Apparent plasma clearance (CL/F) values were calculated as Dose/AUCtau.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hour
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor | Part B - All Tumor Types TMT 0.025 mg/kg/Day | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 3 | 18 | 9 | 15 | 9 | 10 | 10 | 9 | 38 | 1 | 1 | 6 | 20 | 6 | 5 | 21
mL/hour | 2750 (69.4) | 1530 (64.5) | 1240 (25.5) | 2040 (71.5) | 1710 (55.6) | 1910 (47.8) | 1590 (65.3) | 1820 (42.6) | 1750 (51.5) | 2590 | 3770 | 2010 (38.5) | 3540 (54.0) | 3060 (44.9) | 2180 (23.9) | 3810 (49.6)

9. Secondary Outcome: Average Steady State Plasma Concentration (Cavg) of Trametinib When Administered in Combination With Dabrafenib
Description: as for outcome 2
Time Frame: pre dose, 0.5, 1, 2, 3, 4, 6 and 8 hours post trametinib dose on Cycle 1 Day 15. The duration of 1 cycle was 28 days.
Population: All subjects who received at least one dose of trametinib in Part C and D and provided an evaluable PK profile with a value for the outcome measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 1 | 1 | 6 | 20 | 6 | 5 | 21
ng/mL | 12.1 | 13.8 | 9.83 (28.4) | 12.8 (20.0) | 7.76 (23.7) | 9.50 (33.1) | 11.9 (28.4)

10. Secondary Outcome: Incidence of Treatment Emergent Adverse Events in Subjects Treated With Trametinib in Combination With Dabrafenib
Description: as for outcome 1
Time Frame: From the day of the first dose of the combination up to 30 days after the last dose, up to maximum duration of 53 months
Population: All subjects who received at least one dose of any component of the combination in Part C and Part D
Measure: Count of Participants; unit: Participants
Arm/Group | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH
Number analyzed (Participants) | 3 | 9 | 6 | 20 | 10
Participants
  AEs | 3 | 9 | 6 | 20 | 10
  Treatment-related AEs | 3 | 9 | 6 | 20 | 10
  SAEs | 1 | 5 | 2 | 8 | 6
  Treatment-related SAEs | 0 | 2 | 1 | 5 | 3
  Fatal SAEs | 0 | 0 | 0 | 0 | 0
  AEs leading to discontinuation | 0 | 3 | 1 | 5 | 1
  AEs requiring dose interruptions | 1 | 6 | 4 | 16 | 8
  AEs requiring dose reductions | 1 | 3 | 1 | 6 | 1
  AEs requiring dose reductions or interruptions | 1 | 7 | 4 | 16 | 8

11. Secondary Outcome: Best Overall Response (BOR) Based on RECIST v1.1, RANO and Dombi Criteria and as Per Investigator Assessment
Description: Response evaluations were assessed using Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1) for subjects with solid tumors except neuroblastomas, primary central nervous system tumors (gliomas) or plexiform neurofibromas (PNs).
  Response evaluations for subjects with neuroblastomas could have included: measureable disease (by CT/MRI alone) assessed according to RECIST v1.1, evaluable disease assessed for meta-iodobenzylguanidine (MIBG) response, and biochemical (urine HVA/VMA) with bone marrow involvement assessed by Hematoxylin and Eosin staining of bilateral bone marrow biopsies and aspirates.
  Response evaluations for glioma subjects was assessed using Response Assessment in Neuro Oncology (RANO) criteria with solid tumors through MRI scans.
  Response evaluations of PNs were assessed using volumetric determination and Dombi criteria through MRI scans.
  The number of participants in each response category is reported in the table.
Time Frame: From the day of the first dose of any study drug up to the last dose, up to maximum duration of 63 months
Population: All subjects who received at least one dose of trametinib in Part A and Part B or at least one dose of any component of the combination in Part C and Part D
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH
Number analyzed (Participants) | 3 | 19 | 12 | 16 | 11 | 10 | 10 | 10 | 3 | 9 | 6 | 20 | 10
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3
  Partial response (PR) | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 5 | 2 | 3 | 2 | 9 | 3
  Stable disease (SD) | 1 | 2 | 3 | 4 | 1 | 7 | 8 | 4 | 1 | 5 | 1 | 8 | 3
  Progressive disease (PD) | 0 | 0 | 2 | 0 | 5 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Non-CR/Non-PD | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Missing | 2 | 16 | 6 | 10 | 3 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1

12. Secondary Outcome: Objective Response Rate (ORR) Based on RECIST v1.1, RANO and Dombi Criteria and as Per Investigator Assessment
Description: Objective response rate (ORR) was defined as the percentage of subjects with best overall response rate (BOR) with confirmation of complete response (CR) or partial response (PR) according to criteria for a specific disease type, among subjects with disease assessment at baseline. BOR for each subject was determined from the sequence of overall responses according to the rules for RECIST v1.1, RANO and Dombi criteria. ORR was calculated based on the investigator assessment of tumor response data and was based on confirmed responses.
Time Frame: From the day of the first dose of any study drug up to the last dose, up to maximum duration of 63 months
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH
Number analyzed (Participants) | 3 | 19 | 12 | 16 | 11 | 10 | 10 | 10 | 3 | 9 | 6 | 20 | 10
percentage of participants | 0 [0.0 to 70.8] | 5.3 [0.1 to 26.0] | 8.3 [0.2 to 38.5] | 0 [0.0 to 20.6] | 9.1 [0.2 to 41.3] | 30.0 [6.7 to 65.2] | 0 [0.0 to 30.8] | 50.0 [18.7 to 81.3] | 66.7 [9.4 to 99.2] | 33.3 [7.5 to 70.1] | 66.7 [22.3 to 95.7] | 55.0 [31.5 to 76.9] | 60.0 [26.2 to 87.8]

13. Secondary Outcome: Clinical Benefit Rate (CBR) Based on RECIST v1.1, RANO and Dombi Criteria and as Per Investigator Assessment
Description: Clinical Benefit Rate (CBR) was defined as the percentage of subjects with best overall response rate (BOR) with confirmation of complete response (CR), partial response (PR) or stable disease (SD) according to criteria for a specific disease type, among subjects with disease assessment at baseline. BOR for each subject was determined from the sequence of overall responses according to the rules for RECIST v1.1, RANO and Dombi criteria. ORR was calculated based on the investigator assessment of tumor response data and was based on confirmed responses.
Time Frame: From the day of the first dose of any study drug up to the last dose, up to maximum duration of 63 months
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH
Number analyzed (Participants) | 3 | 19 | 12 | 16 | 11 | 10 | 10 | 10 | 3 | 9 | 6 | 20 | 10
percentage of participants | 33.3 [0.8 to 90.6] | 15.8 [3.4 to 39.6] | 33.3 [9.9 to 65.1] | 25.0 [7.3 to 52.4] | 18.2 [2.3 to 51.8] | 100 [69.2 to 100] | 80.0 [44.4 to 97.5] | 90.0 [55.5 to 99.7] | 100 [29.2 to 100] | 88.9 [51.8 to 99.7] | 83.3 [35.9 to 99.6] | 95.0 [75.1 to 99.9] | 90.0 [55.5 to 99.7]

14. Secondary Outcome: Apparent Clearance (CL/F) of Trametinib Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of trametinib can be described using a two-compartment model with dual sequential 1st order absorption (Ka1, Ka2) and 1st order elimination. Apparent clearance (CL/F) of trametinib estimated with the PopPK model is summarized in this record.
Time Frame: as for outcome 4
Population: All subjects who received at least one dose of trametinib in Part A, B, C and D and provided an evaluable PK profile. All trametinib and dabrafenib concentration-time data were combined and included in a population PK analysis that examined the influence of demographics on the PK of study treatment.
Measure: Number; unit: liters/hour
Groups:
- Part A, B, C and D - All Participants With PK Data: Participants in the study (all doses and all tumor types) with available pharmacokinetic data
Arm/Group | Part A, B, C and D - All Participants With PK Data
Number analyzed (Participants) | 133
liters/hour | 5.07

15. Secondary Outcome: Apparent Central Volume (Vc/F) of Trametinib Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of trametinib can be described using a two-compartment model with dual sequential 1st order absorption (Ka1, Ka2) and 1st order elimination. Apparent central volume (Vc/F) of trametinib estimated with the PopPK model is summarized in this record.
Time Frame: as for outcome 4
Population: as for outcome 14
Measure: Number; unit: liters
Arm/Group | Part A, B, C and D - All Participants With PK Data
Number analyzed (Participants) | 133
liters | 184

16. Secondary Outcome: Absorption Rate Constants (Ka1 and Ka2) of Trametinib Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of trametinib can be described using a two-compartment model with dual sequential 1st order absorption (Ka1, Ka2) and 1st order elimination. The absorption rate constants (Ka1 and Ka2) estimated with the PopPK model are summarized in this record.
Time Frame: as for outcome 4
Population: as for outcome 14
Measure: Number; unit: 1/hours
Arm/Group | Part A, B, C and D - All Participants With PK Data
Number analyzed (Participants) | 133
1/hours
  Ka1 | 0.134
  Ka2 | 1.55

17. Secondary Outcome: Significant Covariates Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of trametinib can be described using a two-compartment model with dual sequential 1st order absorption (Ka1, Ka2) and 1st order elimination. Sex and weight are significant covariates on apparent clearance (CL/F), and weight is also a significant covariate on apparent intercompartmental clearance (Q/F). Use of dabrafenib, yes or no, is a covariate on the relative bioavailability of trametinib, reflecting the effect of dabrafenib on the PK of trametinib.
  The estimates of these covariates (effect of weight on CL/F, effect of sex on CL/F, effect of weight on Q/F, effect of combination with dabrafenib on relative bioavailability F1) calculated with the PopPK model are summarized in this record.
Time Frame: as for outcome 4
Population: as for outcome 14
Measure: Number; unit: no units
Arm/Group | Part A, B, C and D - All Participants With PK Data
Number analyzed (Participants) | 133
no units
  Effect of weight on CL/F | 0.788
  Effect of sex on CL/F | 1.24
  Effect of weight on Q/F | 0.679
  Effect of combination with dabrafenib on relative bioavailability F1 | 0.876

18. Secondary Outcome: Trough Concentration (Ctrough) of Dabrafenib When Administered in Combination With Trametinib
Description: Pharmacokinetic (PK) parameters were calculated based on dabrafenib plasma concentrations by using non-compartmental methods. Ctrough is defined as the observed plasma concentration just prior to the beginning of, or at the end, of a dosing interval.
Time Frame: pre dose on Cycle 1 Day 15. The duration of 1 cycle was 28 days.
Population: All subjects who received at least one dose of dabrafenib in Part C and D and provided an evaluable PK profile with a value for the outcome measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 3 | 7 | 6 | 19 | 8 | 6 | 21
ng/mL | 88.9 (99.6) | 28.6 (203.5) | 8.10 (159.6) | 38.2 (130.9) | 11.8 (869.4) | 5.36 (429.6) | 42.7 (137.4)

19. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Dabrafenib When Administered in Combination With Trametinib
Description: Pharmacokinetic (PK) parameters were calculated based on dabrafenib plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed plasma concentration following a dose.
Time Frame: pre dose, 0.5, 1, 2, 3, 4, 6 and 8 hours post dabrafenib dose on Cycle 1 Day 15. The duration of 1 cycle was 28 days.
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 3 | 7 | 6 | 19 | 8 | 6 | 21
ng/mL | 630 (235.2) | 1560 (35.3) | 1440 (43.3) | 1360 (55.6) | 1490 (88.1) | 1840 (35.2) | 1290 (68.7)

20. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Dabrafenib When Administered in Combination With Trametinib
Description: Pharmacokinetic (PK) parameters were calculated based on dabrafenib plasma concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) plasma concentration following a dose.
Time Frame: pre dose, 0.5, 1, 2, 3, 4, 6 and 8 hours post dabrafenib dose on Cycle 1 Day 15. The duration of 1 cycle was 28 days.
Population: as for outcome 18
Measure: Median (Full Range); unit: hours
Arm/Group | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 3 | 7 | 6 | 19 | 8 | 6 | 21
hours | 2.00 [2.00 to 4.00] | 1.00 [1.00 to 2.00] | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00] | 2.00 [1.00 to 3.00]

21. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast) of Dabrafenib When Administered in Combination With Trametinib
Description: Pharmacokinetic (PK) parameters were calculated based on dabrafenib plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for area under the curve calculation.
Time Frame: pre dose, 0.5, 1, 2, 3, 4, 6 and 8 hours post dabrafenib dose on Cycle 1 Day 15. The duration of 1 cycle was 28 days.
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 3 | 7 | 6 | 19 | 8 | 6 | 21
hours*ng/mL | 2560 (157.1) | 4160 (24.6) | 3910 (48.8) | 4030 (46.4) | 3800 (35.4) | 3990 (28.3) | 3950 (46.9)

22. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau at Steady-state (AUCtau) of Dabrafenib When Administered in Combination With Trametinib
Description: Pharmacokinetic (PK) parameters were calculated based on dabrafenib plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for area under the curve calculation. The duration of the dosing interval (tau) was 12 hours for dabrafenib.
Time Frame: pre dose, 0.5, 1, 2, 3, 4, 6 and 8 hours post dabrafenib dose on Cycle 1 Day 15. The duration of 1 cycle was 28 days.
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 3 | 7 | 6 | 19 | 8 | 6 | 21
hours*ng/mL | 2870 (116.6) | 4160 (24.6) | 4040 (47.9) | 4070 (46.7) | 3910 (37.4) | 4150 (30.2) | 3990 (47.3)

23. Secondary Outcome: Apparent Plasma Clearance (CL/F) of Dabrafenib When Administered in Combination With Trametinib
Description: Pharmacokinetic (PK) parameters were calculated based on dabrafenib plasma concentrations by using non-compartmental methods. Apparent plasma clearance (CL/F) values were calculated as Dose/AUCtau.
Time Frame: pre dose, 0.5, 1, 2, 3, 4, 6 and 8 hours post dabrafenib dose on Cycle 1 Day 15. The duration of 1 cycle was 28 days.
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hour
Arm/Group | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 3 | 7 | 6 | 19 | 8 | 6 | 21
mL/hour | 22900 (191.2) | 20400 (45.4) | 10100 (67.0) | 25400 (70.5) | 12500 (63.0) | 10200 (41.6) | 25100 (69.3)

24. Secondary Outcome: Average Steady State Plasma Concentration (Cavg) of Dabrafenib When Administered in Combination With Trametinib
Description: Pharmacokinetic (PK) parameters were calculated based on dabrafenib plasma concentrations by using non-compartmental methods. The average steady state plasma concentration (Cavg) of dabrafenib was calculated as the ratio of area under the curve (AUC)/tau, where tau = 12 h for dabrafenib.
Time Frame: pre dose, 0.5, 1, 2, 3, 4, 6 and 8 hours post dabrafenib dose on Cycle 1 Day 15. The duration of 1 cycle was 28 days.
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH | Part D - All Tumor Types TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - All Tumor Types TMT 0.025 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 3 | 7 | 6 | 19 | 8 | 6 | 21
ng/mL | 239 (116.6) | 347 (24.6) | 337 (47.9) | 339 (46.7) | 326 (37.4) | 346 (30.2) | 332 (47.3)

25. Secondary Outcome: Palatability of Trametinib Oral Solution in Pediatric Subjects Assessed by Palatability Questionnaire
Description: For subjects ≥ 12 years of age who received the trametinib oral solution, the subject completed a form to evaluate the various properties of the solution (e.g., bitterness, sweetness, appearance, texture and overall taste). For subjects < 12 years of age who received the solution, their caregiver (e.g. parent or guardian) evaluated the solution with the child based on verbal and non-verbal feedback. The questionnaire was completed after the first dose of study drug and no later than Day 8 (±3 days). Subjects completed a form for each drug separately if enrolled in Parts C and D.
Time Frame: After the first dose of trametinib oral solution and no later than Day 8 (±3 days)
Population: All subjects who received at least one dose of trametinib oral solution and filled in the palatability questionnaire.
  All palatability questionnaire results were combined and reported based on drug dose to better determine the acceptability and palatability of the formulation.
Measure: Count of Participants; unit: Participants
Groups:
- TMT 0.0125 mg/kg/Day: Participants treated with trametinib oral solution at a dose level of 0.0125 mg/kg/day
- TMT 0.025 mg/kg/Day: Participants treated with trametinib oral solution at a dose level of 0.025 mg/kg/day
- TMT 0.032 mg/kg/Day: Participants treated with trametinib oral solution at a dose level of 0.032 mg/kg/day
- TMT 0.04 mg/kg/Day: Participants treated with trametinib oral solution at a dose level of 0.04 mg/kg/day
Arm/Group | TMT 0.0125 mg/kg/Day | TMT 0.025 mg/kg/Day | TMT 0.032 mg/kg/Day | TMT 0.04 mg/kg/Day
Number analyzed (Participants) | 2 | 29 | 21 | 4
Participants
  Was the medicine difficult to mix?: Yes | 0 | 1 | 1 | 0
  Was the medicine difficult to mix?: No | 2 | 26 | 19 | 4
  Was the medicine difficult to mix?: missing | 0 | 2 | 1 | 0
  Was the medicine difficult to measure?: Yes | 0 | 0 | 2 | 0
  Was the medicine difficult to measure?: No | 2 | 29 | 18 | 4
  Was the medicine difficult to measure?: missing | 0 | 0 | 1 | 0
  Was the medicine difficult to administer?: Yes | 0 | 5 | 5 | 1
  Was the medicine difficult to administer?: No | 2 | 24 | 15 | 3
  Was the medicine difficult to administer?: missing | 0 | 0 | 1 | 0
  Did the subject like the taste of the medicine?: Yes | 2 | 8 | 6 | 2
  Did the subject like the taste of the medicine?: No | 0 | 16 | 13 | 1
  Did the subject like the taste of the medicine?: missing | 0 | 5 | 2 | 1
  Did the subject have difficulty in taking the medicine?: Yes | 0 | 6 | 7 | 1
  Did the subject have difficulty in taking the medicine?: No | 2 | 19 | 13 | 3
  Did the subject have difficulty in taking the medicine?: missing | 0 | 4 | 1 | 0
  Did the subject resist taking the medicine?: Yes | 0 | 7 | 6 | 1
  Did the subject resist taking the medicine?: No | 2 | 18 | 14 | 3
  Did the subject resist taking the medicine?: missing | 0 | 4 | 1 | 0
  Was the medicine bitter?: Yes | 0 | 3 | 0 | 0
  Was the medicine bitter?: No | 0 | 2 | 1 | 0
  Was the medicine bitter?: missing | 2 | 24 | 20 | 4
  Was the medicine sweet?: Yes | 0 | 2 | 1 | 0
  Was the medicine sweet?: No | 0 | 3 | 0 | 0
  Was the medicine sweet?: missing | 2 | 24 | 20 | 4
  Was the medicine sour?: Yes | 0 | 2 | 0 | 0
  Was the medicine sour?: No | 0 | 3 | 1 | 0
  Was the medicine sour?: missing | 2 | 24 | 20 | 4
  Was the medicine gritty?: Yes | 0 | 1 | 0 | 0
  Was the medicine gritty?: No | 0 | 4 | 1 | 0
  Was the medicine gritty?: missing | 2 | 24 | 20 | 4
  Was the medicine difficult to swallow?: Yes | 0 | 1 | 0 | 0
  Was the medicine difficult to swallow?: No | 0 | 5 | 1 | 0
  Was the medicine difficult to swallow?: missing | 2 | 23 | 20 | 4

26. Secondary Outcome: Palatability of Dabrafenib Oral Suspension in Pediatric Subjects Assessed by Palatability Questionnaire
Description: For subjects ≥ 12 years of age who received the dabrafenib suspension, the subject completed a form to evaluate the various properties of the suspension (e.g., bitterness, sweetness, appearance, texture and overall taste). For subjects < 12 years of age who received the suspension, their caregiver (e.g. parent or guardian) evaluated the suspension with the child based on verbal and non-verbal feedback. The questionnaire was completed after the first dose of study drug and no later than Day 8 (±3 days). Subjects completed a form for each drug separately if enrolled in Parts C and D.
Time Frame: After the first dose of dabrafenib oral suspension and no later than Day 8 (±3 days)
Population: All subjects who received at least one dose of dabrafenib oral suspension and filled in the palatability questionnaire.
  All palatability questionnaire results were combined and reported based on drug dose to better determine the acceptability and palatability of the formulation. There were no results available for participants who received 50% of the RP2D of dabrafenib monotherapy in combination with trametinib because the participants did not fill in the questionnaire.
Measure: Count of Participants; unit: Participants
Groups:
- TMT 0.025 mg/kg/Day + 50% DRB RP2D: Participants treated with a combination therapy of trametinib (0.025 mg/kg/day) plus 50% of the RP2D of dabrafenib monotherapy (oral suspension formulation)
- TMT 0.025 mg/kg/Day + 100% DRB RP2D: Participants treated with a combination therapy of trametinib (0.025 mg/kg/day) plus 100% of the RP2D of dabrafenib monotherapy (oral suspension formulation)
- TMT 0.032 mg/kg/Day + 100% DRB RP2D: Participants treated with a combination therapy of trametinib (0.032 mg/kg/day) plus 100% of the RP2D of dabrafenib monotherapy (oral suspension formulation)
Arm/Group | TMT 0.025 mg/kg/Day + 50% DRB RP2D | TMT 0.025 mg/kg/Day + 100% DRB RP2D | TMT 0.032 mg/kg/Day + 100% DRB RP2D
Number analyzed (Participants) | 0 | 4 | 6
Participants
  Was the medicine difficult to mix?: Yes |  | 0 | 1
  Was the medicine difficult to mix?: No |  | 4 | 5
  Was the medicine difficult to mix?: missing |  | 0 | 0
  Was the medicine difficult to measure?: Yes |  | 0 | 1
  Was the medicine difficult to measure?: No |  | 4 | 5
  Was the medicine difficult to measure?: missing |  | 0 | 0
  Was the medicine difficult to administer?: Yes |  | 0 | 1
  Was the medicine difficult to administer?: No |  | 4 | 5
  Was the medicine difficult to administer?: missing |  | 0 | 0
  Did the subject like the taste of the medicine?: Yes |  | 0 | 4
  Did the subject like the taste of the medicine?: No |  | 1 | 2
  Did the subject like the taste of the medicine?: missing |  | 3 | 0
  Did the subject have difficulty in taking the medicine?: Yes |  | 0 | 2
  Did the subject have difficulty in taking the medicine?: No |  | 1 | 4
  Did the subject have difficulty in taking the medicine?: missing |  | 3 | 0
  Did the subject resist taking the medicine?: Yes |  | 0 | 4
  Did the subject resist taking the medicine?: No |  | 1 | 2
  Did the subject resist taking the medicine?: missing |  | 3 | 0
  Was the medicine bitter?: Yes |  | 1 | 0
  Was the medicine bitter?: No |  | 2 | 0
  Was the medicine bitter?: missing |  | 1 | 6
  Was the medicine sweet?: Yes |  | 0 | 0
  Was the medicine sweet?: No |  | 3 | 0
  Was the medicine sweet?: missing |  | 1 | 6
  Was the medicine sour?: Yes |  | 2 | 0
  Was the medicine sour?: No |  | 1 | 0
  Was the medicine sour?: missing |  | 1 | 6
  Was the medicine gritty?: Yes |  | 1 | 0
  Was the medicine gritty?: No |  | 2 | 0
  Was the medicine gritty?: missing |  | 1 | 6
  Was the medicine difficult to swallow?: Yes |  | 0 | 0
  Was the medicine difficult to swallow?: No |  | 3 | 0
  Was the medicine difficult to swallow?: missing |  | 1 | 6

ADVERSE EVENTS:
Time Frame: From the day of the first dose of any study drug up to 30 days after the last dose, up to maximum duration of 64 months.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Arm/Group | Part A - TMT 0.0125 mg/kg/Day | Part A - TMT 0.025 mg/kg/Day | Part A - TMT 0.032 mg/kg/Day | Part A - TMT 0.04 mg/kg/Day | Part B - Neuroblastoma | Part B - LGG Fusion | Part B - NF-1 With PN | Part B - BRAF V600 Mutant Solid Tumor | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D | Part D - LGG | Part D - LCH
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/19 | 0/12 | 0/16 | 0/11 | 0/10 | 0/10 | 0/10 | 0/3 | 0/9 | 0/6 | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/3 | 8/19 | 3/12 | 11/16 | 6/11 | 6/10 | 6/10 | 5/10 | 1/3 | 5/9 | 2/6 | 8/20 | 6/10
Other Adverse Events (participants affected / at risk) | 3/3 | 19/19 | 12/12 | 16/16 | 11/11 | 10/10 | 10/10 | 10/10 | 3/3 | 9/9 | 6/6 | 20/20 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - TMT 0.0125 mg/kg/Day (N=3) | Part A - TMT 0.025 mg/kg/Day (N=19) | Part A - TMT 0.032 mg/kg/Day (N=12) | Part A - TMT 0.04 mg/kg/Day (N=16) | Part B - Neuroblastoma (N=11) | Part B - LGG Fusion (N=10) | Part B - NF-1 With PN (N=10) | Part B - BRAF V600 Mutant Solid Tumor (N=10) | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D (N=3) | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D (N=9) | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D (N=6) | Part D - LGG (N=20) | Part D - LCH (N=10)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 1 | 2 | 0 | 2 | 2 | 0 | 3 | 1 | 4 | 4
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Enterobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood culture positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal tube insertion (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - TMT 0.0125 mg/kg/Day (N=3) | Part A - TMT 0.025 mg/kg/Day (N=19) | Part A - TMT 0.032 mg/kg/Day (N=12) | Part A - TMT 0.04 mg/kg/Day (N=16) | Part B - Neuroblastoma (N=11) | Part B - LGG Fusion (N=10) | Part B - NF-1 With PN (N=10) | Part B - BRAF V600 Mutant Solid Tumor (N=10) | Part C - TMT 0.025 mg/kg/Day + 50% DRB RP2D (N=3) | Part C - TMT 0.025 mg/kg/Day + 100% DRB RP2D (N=9) | Part C - TMT 0.032 mg/kg/Day + 100% DRB RP2D (N=6) | Part D - LGG (N=20) | Part D - LCH (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 9 | 6 | 7 | 6 | 3 | 4 | 5 | 0 | 4 | 1 | 4 | 2
Bone marrow oedema (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypochromasia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve disease (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 5 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 3 | 0 | 2 | 1
Systolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Growth hormone deficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypogonadism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Precocious puberty (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Amblyopia (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Astigmatism (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bell's phenomenon (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyschromatopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid margin crusting (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gaze palsy (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heterophoria (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mydriasis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Ocular hypertension (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Optic disc disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Optic disc haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pupillary reflex impaired (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trichomegaly (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 8 | 7 | 5 | 1 | 5 | 1 | 2 | 0 | 3 | 2 | 6 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal rash (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angular cheilitis (Gastrointestinal disorders) | 0 | 4 | 1 | 2 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 2 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 3 | 6 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 8 | 6 | 3 | 4 | 5 | 2 | 6 | 1 | 2 | 1 | 5 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 17 | 10 | 9 | 6 | 6 | 5 | 6 | 2 | 3 | 3 | 7 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 0 | 3 | 0 | 2 | 0 | 1 | 0 | 1 | 0
Lip haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 6 | 1 | 4 | 3 | 2 | 3 | 3 | 0 | 4 | 1 | 8 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 3 | 3 | 2 | 1 | 4 | 3 | 2 | 0 | 2 | 0 | 1 | 0
Teething (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 13 | 9 | 6 | 3 | 3 | 3 | 6 | 1 | 4 | 4 | 9 | 7
Asthenia (General disorders) | 0 | 4 | 0 | 4 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Catheter site hypersensitivity (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 3 | 0
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 10 | 9 | 4 | 1 | 1 | 0 | 6 | 2 | 4 | 1 | 9 | 4
Feeling cold (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Granuloma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 2 | 3
Localised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Mucosal inflammation (General disorders) | 0 | 4 | 1 | 1 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1
Pain (General disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 11 | 8 | 10 | 5 | 5 | 6 | 4 | 0 | 7 | 4 | 15 | 8
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xerosis (General disorders) | 0 | 4 | 2 | 2 | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 2 | 1 | 4 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coxsackie viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 6 | 3 | 4 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 3 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes dermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected bite (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymph gland infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal vestibulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 3 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 2
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Paronychia (Infections and infestations) | 0 | 16 | 10 | 12 | 0 | 4 | 7 | 7 | 2 | 1 | 1 | 6 | 1
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pustule (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 1 | 5 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 4 | 0 | 2 | 0 | 2 | 3 | 1 | 0 | 2 | 0 | 2 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Skin bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 4 | 2 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tinea capitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea faciei (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 6 | 3 | 1 | 0 | 0 | 3 | 3 | 0 | 2 | 1 | 6 | 4
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 4 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Incision site pruritus (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Stoma site hypergranulation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Venomous sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 3 | 1 | 5 | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 3 | 0
Albumin urine present (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anion gap decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 8 | 4 | 7 | 3 | 1 | 1 | 6 | 1 | 3 | 3 | 5 | 1
Bacterial test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 5 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 2 | 2 | 2 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bicarbonate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood chloride increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 3 | 1 | 2 | 5 | 1 | 0 | 1 | 0 | 2 | 2 | 0 | 2
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urea decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body temperature fluctuation (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram ST-T segment abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave amplitude decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
End-tidal CO2 decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 2 | 1 | 2 | 2 | 3 | 1
Grip strength decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lung diffusion test decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 2 | 2 | 1 | 2 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 1
Lymphocyte count increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte percentage decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 3 | 0 | 3 | 5
Neutrophil percentage increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nitrite urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Protein total decreased (Investigations) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Protein urine (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Red blood cells urine (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Specific gravity urine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine ketone body present (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 5 | 3 | 0 | 2 | 3 | 0 | 1 | 1 | 1 | 2 | 5 | 1
White blood cell count decreased (Investigations) | 0 | 2 | 3 | 4 | 3 | 1 | 0 | 0 | 0 | 2 | 0 | 3 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
pH urine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 11 | 4 | 5 | 1 | 3 | 2 | 3 | 0 | 1 | 0 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 3 | 4 | 3 | 2 | 1 | 2 | 0 | 3 | 0 | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 5 | 1 | 2 | 1 | 1 | 0 | 3 | 0 | 2 | 1 | 2 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 5 | 6 | 4 | 4 | 3 | 1 | 3 | 0 | 4 | 2 | 3 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 5 | 3 | 2 | 1 | 1 | 2 | 0 | 4 | 0 | 2 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 2 | 4 | 1 | 0 | 1 | 1 | 0 | 3 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 2 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 3 | 1 | 0 | 2 | 0 | 1 | 1 | 3 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salt craving (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2 | 3 | 1 | 2 | 0 | 1 | 1 | 4 | 0 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 4 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 7 | 3 | 3 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 3 | 4
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toe walking (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allodynia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aura (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 4 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 11 | 3 | 5 | 1 | 4 | 4 | 3 | 1 | 4 | 1 | 9 | 2
Horner's syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Movement disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dyssomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enuresis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 4 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2
Irritability (Psychiatric disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Albuminuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crystalluria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 4 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 4 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 4 | 3 | 2 | 3 | 2 | 0 | 3 | 0 | 3 | 2 | 1 | 0
Urethritis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perineal rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 6 | 4 | 2 | 4 | 5 | 4 | 1 | 4 | 1 | 8 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 4 | 8 | 2 | 2 | 1 | 2 | 1 | 2 | 0 | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 2 | 1 | 5 | 3
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal odour (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 2 | 0 | 1 | 1 | 3 | 1 | 3 | 0 | 3 | 2
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4 | 1 | 1 | 2 | 1 | 1 | 0 | 3 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 7 | 4 | 6 | 1 | 5 | 4 | 3 | 0 | 1 | 1 | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 6 | 4 | 10 | 1 | 4 | 3 | 4 | 2 | 4 | 1 | 8 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 12 | 10 | 6 | 4 | 7 | 5 | 6 | 2 | 5 | 3 | 8 | 5
Eczema (Skin and subcutaneous tissue disorders) | 1 | 8 | 5 | 9 | 2 | 5 | 1 | 1 | 1 | 0 | 0 | 3 | 2
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 5 | 1 | 5 | 2 | 0 | 0 | 3 | 0 | 1 | 0 | 2 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Plantar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 5 | 1 | 4 | 2 | 1 | 1 | 3 | 0 | 2 | 0 | 3 | 3
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 9 | 5 | 8 | 4 | 5 | 6 | 2 | 3 | 6 | 2 | 3 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 3 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3 | 4 | 4 | 2 | 4 | 2 | 3 | 1 | 0 | 2 | 6 | 5
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 4 | 3 | 3 | 0 | 2 | 0 | 4 | 0 | 1 | 0 | 2 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Skin fragility (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0
Central venous catheter removal (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tonsillectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 3 | 3 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT02124772/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT02124772/SAP_001.pdf